CLINICAL TRIAL: NCT02013219
Title: A Phase 1b Study of the Safety and Pharmacology of Atezolizumab (Anti-PD-L1 Antibody) Administered With Erlotinib or Alectinib in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: A Phase 1b Study of Atezolizumab in Combination With Erlotinib or Alectinib in Participants With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WP29158; 2013-004382-13 (EudraCT Number)
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib; atezolizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stage 1: Alectinib and Atezolizumab (Experimental): In Stage 1, starting dose of atezolizumab will be 1200 mg IV q3w administered on Day 8 of Cycle 1 and on Day 1 (21-day cycle) of each cycle thereafter along with alectinib at a starting dose of 600 mg PO BID for 28 consecutive days during Cycle 1 and on Days 1-21 of each cycle thereafter; unless maximum tolerable dose (MTD) is exceeded. The combination will be given to treatment-naive participants with ALK-positive, locally advanced or metastatic NSCLC.
  Interventions: Drug: Alectinib; Drug: Atezolizumab
- Stage 1: Erlotinib and Atezolizumab (Experimental): In Stage 1, starting dose of atezolizumab will be 1200 mg IV q3w administered on Day 8 of Cycle 1 and on Day 1 (21-day cycles) of each cycle thereafter along with erlotinib at a starting dose of 150 mg PO QD, for 28 consecutive days during Cycle 1 and on Days 1-21 of each cycle thereafter; unless MTD is exceeded. The combination will be given to participants with EGFR TKI treatment-naive, locally advanced or metastatic NSCLC.
  Interventions: Drug: Atezolizumab; Drug: Erlotinib
- Stage 2: Alectinib and Atezolizumab (Experimental): In Stage 2, participants received the RP2D on the basis of the MTD or maximum allowed dose (MAD) of the combination treatment established in Stage 1. Treatment-naive participants with ALK-positive, locally advanced or metastatic NSCLC will be included.
  Interventions: Drug: Alectinib; Drug: Atezolizumab
- Stage 2: Erlotinib and Atezolizumab (Experimental): In Stage 2, participants received the RP2D on the basis of the MTD or MAD of the combination treatment established in Stage 1. Previously untreated (or with one prior treatment that was not an EGFR TKI), EGFR mutation positive, locally advanced or metastatic NSCLC participants will be included.
  Interventions: Drug: Atezolizumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Alectinib — Participants will receive 600 mg PO alectinib BID for 28 consecutive days during Cycle 1 and on Days 1-21 of each cycle thereafter (21-day cycles from Cycle 2 onwards) in Stage 1 and RP2D PO BID in Stage 2.
  Other Names: Alecensa
  Arms: Stage 1: Alectinib and Atezolizumab; Stage 2: Alectinib and Atezolizumab
Drug: Atezolizumab — Participants will receive 1200 mg atezolizumab IV infusion q3w on Day 8 of Cycle 1 and on Day 1 of each cycle thereafter in Stage 1 and in Stage 2.
  Other Names: TECENTRIQ; MPDL3280A
Drug: Erlotinib — Participants will receive 150 mg erlotinib PO QD for 28 consecutive days during Cycle 1 and on Days 1-21 of each cycle thereafter in Stage 1 (21-day cycles from Cycle 2 onwards) and RP2D PO QD in Stage 2.
  Other Names: Tarceva
  Arms: Stage 1: Erlotinib and Atezolizumab; Stage 2: Erlotinib and Atezolizumab

SUMMARY:
This open-label, multicenter study will assess the safety, tolerability, and pharmacokinetics of intravenous (IV) dosing of atezolizumab in combination with oral erlotinib or alectinib in participants with NSCLC.

This study has two stages. In the erlotinib group, the combination treatment will be given to participants with epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI)-treatment-naive, advanced (nonresectable) NSCLC in a safety-evaluation stage and to participants with previously untreated EGFR mutation-positive, advanced NSCLC in an expansion stage (Stage 2). In the alectinib group, for both the safety-evaluation and expansion stages (Stages 1 and 2), the combination will be given to participants who are treatment-naive with anaplastic lymphoma kinase (ALK)-positive advanced NSCLC.

In Stage 1, erlotinib will be given at a starting dose of 150 milligrams (mg) by mouth (PO) once daily (QD) and the starting dose of alectinib will be 600 mg twice daily (BID), for 28 consecutive days during Cycle 1 and on Days 1 through 21 of each cycle thereafter. The starting dose of atezolizumab will be 1200 mg, administered every 3 weeks (q3W) starting on Day 8 of Cycle 1. If the starting regimen for a combination treatment is not tolerated, alternative doses and/or schedules of erlotinib and atezolizumab or alectinib and atezolizumab may be tested to determine potential recommended Phase 2 dose (RP2D) for that combination treatment. In Stage 2, a potential RP2D and schedule for each combination treatment will be investigated in an expansion cohort.

For both stages, continuation of treatment beyond Cycle 1 will be at the discretion of the treating investigator. Study treatment will be discontinued in participants who experience disease progression or unacceptable toxicity, are not compliant with the study protocol, or, in their opinion or in the opinion of the investigator, are not benefiting from study treatment. However, in the absence of unacceptable toxicity, participants with second-line or greater NSCLC who are still receiving atezolizumab at the time of radiographic disease progression may be permitted to continue study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, locally advanced or metastatic NSCLC.
* Participants in Stage 1 (Safety Evaluation) receiving erlotinib: No limit to the number of prior therapies (except for EGFR TKIs).
* Participants in Stage 2 (Expansion) receiving erlotinib: i) sensitizing mutation in the EGFR gene and ii) consent to collection of tumor tissue samples before, during, and after treatment for biopsy and PD biomarker analyses.
* Participants receiving alectinib in either Stage 1 or Stage 2: must be ALK positive as assessed by Food and Drug Administration (FDA) approved test and must not have received prior treatment for their advanced NSCLC.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 12 weeks.
* Measurable disease, as defined by RECIST Version 1.1 (v1.1).
* Adequate hematologic and end-organ function.
* Use of highly effective contraception (as defined by protocol) and until 5 months after the last dose of atezolizumab and for 3 months after the last dose of alectinib or for 2 weeks after the last dose of erlotinib, whichever is longer; Males must also refrain from sperm donatation during this same time period. Participants must not be pregnant or breastfeeding.
* Archival tumor tissue specimen meeting protocol specifications or the participant will be offered the option of a pre-treatment biopsy to obtain adequate tissue sample.

Exclusion Criteria:

* For participants receiving erlotinib group: prior treatment with any EGFR mutant-targeting TKI
* Any approved anticancer therapy, including chemotherapy, or hormonal therapy (except hormone-replacement therapy or oral contraceptives) within 3 weeks of first dose.
* Treatment with any other test drug or participation in another clinical trial within 28 days of enrollment.
* Known symptomatic central nervous system (CNS) metastases. Participants with a history of treated or untreated asymptomatic CNS metastases may be eligible.
* Leptomeningeal disease.
* Uncontrolled tumor-related pain.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage at least once monthly.
* High levels of calcium requiring bisphosphonate therapy or denosumab.
* Malignancies other than NSCLC within 5 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death (such as adequately treated carcinoma in-situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ).
* History of severe allergic, anaphylactic, or other reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation.
* History of autoimmune disease.
* Participants with prior bone marrow or solid organ transplantation.
* History of lung inflammation or disease.
* Serum albumin less than (<) 2.5 grams per deciliter (g/dL).
* Positive for Human Immunodeficiency Virus (HIV).
* Liver disease.
* Current or active tuberculosis, hepatitis B, or hepatitis C.
* Participants with past or resolved hepatitis B virus (HBV) infection are eligible; participants positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV Riboxy Nucleic Acid (RNA).
* Signs or symptoms of infection within 2 weeks prior to first dosing.
* Received therapeutic oral or IV antibiotics within 2 weeks prior to first dosing.
* Significant cardiovascular disease.
* Major surgical procedure other than for diagnosis within 28 days prior to first dosing or during the course of the study.
* Administration of a live, attenuated vaccine within 4 weeks before first dosing or during the study.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that may reasonably prevent the participant from participating.
* Hypersensitivity to erlotinib or alectinib or to any of the excipients.
* Any significant ophthalmologic abnormality. The use of contact lenses is not recommended during the study.
* For participants receiving alectinib: baseline Fridericias corrected QT interval (QTcF) greater than (>) 470 milliseconds (ms) or symptomatic bradycardia.
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies.
* Treatment with systemic immunostimulatory agents within 6 weeks or five half-lives of the drug, whichever is shorter, prior to first dosing.
* Treatment with systemic immunosuppressive medications within 2 weeks prior to first dosing (inhaled corticosteroids and mineralocorticoids are allowed).
* Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication are elgible for study after discussion and approval by the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | 28 days
Recommended Phase II Dose (RP2D) of Atezolizumab and Erlotinib | 28 days
Recommended RP2D of Atezolizumab and Alectinib | 28 days

SECONDARY OUTCOMES:
Minimum Plasma Concentration (Cmin) of Alectinib and Major Metabolites, as Appropriate | Pre-dose (0 hour) on Day 1 of Cycles 1-4, Day 8 of Cycle 1 (Cycle 1 =28 days; Cycle 2 onwards=21 days)
Progression-Free Survival (PFS) as Assessed Using the Response Evaluation Criteria in Solid Tumors (RECIST) | First dose of study treatment up to disease progression or death from any cause (up to approximately 6 years)
Overall Survival | First dose of study treatment up to death from any cause during the study (up to approximately 6 years)
Percentage of Participants with Objective Response (Complete Response [CR] or Partial Response [PR]) Using RECIST | Baseline up to disease progression or death from any cause (up to approximately 6 years)
Percentage of Participants with Adverse Events | Baseline up to approximately 6 years
Percentage of Participants with Anti-Drug Antibodies (ADAs) Against Atezolizumab | Baseline up to approximately 6 years
Maximum Serum Concentration (Cmax) of Atezolizumab | Day 1 of Cycles 1-4, Day 8 of Cycle 1 (Cycle 1 =21 days; Cycle 2 onwards=28 days)
Minimum Serum Concentration (Cmin) of Atezolizumab | Pre-dose (0 hour) on Day 1 of Cycles 1, 2, 3, 4, 6, and 8 and at study termination (up to approximately 5 years; Cycle 1=21 days; Cycle 2 onwards=28 days)
Maximum Plasma Concentration (Cmax) of Erlotinib | Day 1 of Cycles 1-4, Day 8 of Cycle 1 (Cycle 1 =21 days; Cycle 2 onwards=28 days)
Minimum Plasma Concentration (Cmin) of Erlotinib | Pre-dose (0 hour) on Day 1 of Cycles 1-4, Day 8 of Cycle 1 (Cycle 1 =21 days; Cycle 2 onwards=28 days)
Maximum Plasma Concentration (Cmax) of Alectinib and Major Metabolites, as Appropriate | Day 1 of Cycles 1-4, Day 8 of Cycle 1 (Cycle 1 =21 days; Cycle 2 onwards=28 days)
Duration of Objective Response as Assessed Using RECIST | First occurrence of a documented objective response up to disease progression or death from any cause (up to approximately 6 years)
Percentage of Participants with Best Overall Response | Baseline up to disease progression or death from any cause (up to approximately 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- United States (10):
  - UC Irvine Medical Center, Orange, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Florida Hospital Cancer Inst, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital;Hematology/ Oncology, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr; Neurology/MS Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center; Department of Oncology, Detroit, Michigan
  - Memorial Sloan Kettering - Basking Ridge, New York, New York
  - Case Western Reserve University; Medicine-Hematology and Oncology, Cleveland, Ohio
- Institut Gustave Roussy, Villejuif, France
- The Chinese University of Hong Kong, Shatin, Hong Kong
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (2):
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Queen Mary University of London, London, United Kingdom